CLINICAL TRIAL: NCT04094610
Title: A Phase 1/2, Open-Label, Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity Study of Repotrectinib in Pediatric and Young Adult Subjects With Advanced or Metastatic Malignancies Harboring ALK, ROS1, NTRK1-3 Alterations
Brief Title: A Study of Repotrectinib in Pediatric and Young Adult Subjects Harboring ALK, ROS1, OR NTRK1-3 Alterations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Turning Point Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA127-1029; CA127-1029 (Other: BMS Protocol ID); TPX-0005-07 (Other: Turning Point Therapeutics Protocol ID)
Expanded Access: NCT05926232 (Available)
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors; Lymphoma; Primary CNS Tumors
Keywords: ALK; ROS1; NTRK1-3; Primary CNS tumor; anaplastic large cell lymphoma; metastatic solid tumor; advanced solid tumor; sarcoma; infantile fibrosarcoma; glioblastoma; soft tissue schwannoma; solitary fibrous tumor; glioma; inflammatory myofibroblastic tumor; pediatric
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Neoplasm Metastasis; Sarcoma; Glioblastoma; Solitary Fibrous Tumors; Glioma; Granuloma, Plasma Cell | interventions — repotrectinib; Capsules; Suspensions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Repotrectinib (TPX-0005) (Experimental): Phase 1
  Oral repotrectinib (TPX-0005):
  Safety and tolerability at different dose levels
  Phase 2
  Oral repotrectinib (TPX-0005): 3 cohorts
  Cohort 1: TKI-naive NTRK fusion Cohort 2: Prior TKI NTRK fusion Cohort 3: ROS1 gene fusions or other ROS1 aberrations
  Interventions: Drug: Oral repotrectinib (TPX-0005)

INTERVENTIONS:
Drug: Oral repotrectinib (TPX-0005) — Oral repotrectinib (TPX-0005)
  Other Names: Oral repotrectinib (TPX-0005) capsules; Oral repotrectinib (TPX-0005) oral suspension; repotrectinib

SUMMARY:
Phase 1 will evaluate the safety and tolerability at different dose levels of repotrectinib in pediatric and young adult subjects with advanced or metastatic malignancies harboring anaplastic lymphoma kinase (ALK), receptor tyrosine kinase encoded by the gene ROS1 (ROS1), or neurotrophic receptor kinase genes encoding TRK kinase family (NTRK1-3) alterations to estimate the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD) and select the Pediatric Recommended Phase 2 Dose (RP2D).

Phase 2 will determine the anti-tumor activity of repotrectinib in pediatric and young adult subjects with advanced or metastatic malignancies harboring ROS1 or NTRK1-3 alterations.

DETAILED DESCRIPTION:
Enrollment of subjects into Phase 1 will proceed concurrently by age as follows:

* Subjects <12 years old will initially be enrolled in the Phase 1 part to determine the pediatric RP2D for this age group; once the pediatric RP2D is determined, subjects age <12 years old may be enrolled into the Phase 2 part of the study.
* Subjects 12 to 25 years old will be directly enrolled into the Phase 2 part concurrent with Phase 1 enrollment.

Phase 1:

Approximately 12 pediatric subjects with locally advanced or metastatic solid tumors, including a primary central nervous system (CNS) tumor, or anaplastic large cell lymphoma (ALCL), with disease progression or who are non-responsive or intolerant to available therapies and for which no standard or available curative therapy exists.

Phase 2:

Subjects will be enrolled in one of 3 cohorts as follows:

Cohort 1: approximately 10-20 subjects with solid tumors characterized by NTRK fusion, TRK tyrosine kinase inhibitor (TKI)-naïve, and centrally confirmed measurable disease at baseline.

Cohort 2: approximately 23 subjects with solid tumors characterized by NTRK fusion, TRK TKI-pretreated, and centrally confirmed measurable disease at baseline.

Cohort 3: approximately 20 subjects with solid tumors or ALCL characterized by other ALK/ROS1/NTRK alterations or NTRK fusions without centrally confirmed measurable disease not otherwise eligible for Cohort 1 or 2. As of the current protocol amendment, only patients with ROS1 alterations will be enrolled to this cohort.

ELIGIBILITY:
Key Inclusion Criteria:

1. Documented genetic ROS1 point mutation, fusion, or amplification or NTRK1-3 fusion as identified by local testing in a Clinical Laboratory Improvement Amendments (CLIA) laboratory in the US or equivalently accredited diagnostic lab outside the United States (US) is required.
2. Phase 1: Age <12 years; Phase 2: Age 12- 25 years
3. Prior cytotoxic chemotherapy is allowed.
4. Prior immunotherapy is allowed.
5. Resolution of all acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Grade less than or equal to 1.
6. All subjects must have measurable disease by RECIST v1.1 or Response Assessment in Neuro-Oncology (RANO) criteria at time of enrollment.
7. Subjects with a primary CNS tumor or CNS metastases must be neurologically stable on a stable or decreasing dose of steroids for at least 7 days prior to enrollment.
8. Subjects must have a Lansky (< 16 years) or Karnofsky (≥ 16 years) score of at least 50.
9. Life expectancy greater than or equal to 12 weeks, in the investigator's opinion.
10. Adequate hematologic, renal and hepatic function.

Phase 2 Inclusion Criteria:

1. Cohort Specific Inclusion Criteria:

   * Cohort 1: Subjects with NTRK fusion gene positive (NTRK+) advanced solid tumors (including primary CNS tumors), that are tropomyosin receptor kinase (TRK) TKI naïve;
   * Cohort 2: subjects with NTRK+ advanced solid tumors (including primary CNS tumors), that are TRK TKI pre-treated;
   * Cohort 3: subjects with advanced solid tumors with ROS1 gene fusions or other ROS1 aberrations (including amplifications and point mutations) with measurable disease.
2. Subjects in Cohorts 1 and 2 must have prospectively confirmed measurable disease by BICR prior to enrollment.

Key Exclusion Criteria (Phase 1 and Phase 2):

1. Subjects with neuroblastoma with only bone marrow disease evaluable by bone marrow aspiration only.
2. Major surgery within 14 days (2 weeks) of start of repotrectinib treatment. Central venous access (Broviac, Mediport, etc.) placement does not meet criteria for major surgery.
3. Known active infections requiring ongoing treatment (bacterial, fungal, viral including HIV positivity).
4. Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact drug absorption.
5. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (ECG interval measured from the onset of the QRS complex to the end of the T wave) for heart rate (QTc) > 480 msec obtained from three ECGs, using the screening clinic ECG machine-derived QTc value
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, second degree heart block, PR interval > 250 msec)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval
6. Peripheral neuropathy of CTCAE ≥grade 2.
7. Subjects being treated with or anticipating the need for treatment with strong CYP3A4 inhibitors or inducers.
8. Any potential allergies to repotrectinib and/or its excipients.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLTs) (Phase 1) | Within 28 days of the first repotrectinib dose
  Define the dose limiting toxicities (DLTs) (Phase 1)
Pediatric Recommended Phase 2 Dose (RP2D) (Phase 1) | Within 28 days of the last patient dosed in escalation
  To determine the pediatric RP2D (Phase 1)
Overall Response Rate (ORR) (Phase 2) | Two to three years after first dose of repotrectinib
  To determine the confirmed ORR of repotrectinib (TPX-0005) as assessed by Blinded Independent Central Review (Phase 2)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) (Phase 1) | Approximately three years
  To determine the overall response rate (ORR) by Blinded Independent Central Review (BICR) (Phase 1)
Clinical Benefit Rate (CBR) (Phase 1 and Phase 2) | Approximately three years
  To determine the CBR of repotrectinib (TPX-0005) (Phase 1 and Phase 2)
Time to response (TTR) (Phase 1 and Phase 2) | Approximately three years
  To determine the TTR of reprotrectinib (TPX-005) (Phase 1 and Phase 2)
Duration of response (DOR) (Phase 1 and Phase 2) | Approximately three years
  To determine the DOR of repotrectinib (TPX-0005) (Phase 1 and Phase 2)
Intracranial objective response rate (IC-ORR) (Phase 1 and Phase 2) | Approximately three years
  To determine the IC-ORR of repotrectinib (TPX-005) (Phase 1 and Phase 2)
Central Nervous System Progression-Free Survival (CNS-PFS) (Phase 2) | Approximately three years
  CNS-PFS in subjects with measurable brain metastases (Phase 2)
Progression-free survival (PFS) (Phase 2) | Approximately three years
  To determine the PFS (Phase 2)
Overall survival (OS) (Phase 2) | Approximately three years
  To determine the OS (Phase 2)
Maximum concentration of repotrectinib in plasma (Cmax) | Pre-dose and up to 24 hours post-dose on Day 1 and Day 15 in Cycle 1 (each cycle is 28 days)
  To determine the Cmax
Area under the concentration versus time curve of repotrectinib in plasma (AUC) | Pre-dose and up to 24 hours post-dose on Day 1 and Day 15 in Cycle 1 (each cycle is 28 days)
  To determine the AUC

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (68):
- United States (20):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at Los Angeles, Los Angeles, California
  - Children's Hospital Colorado - Anschutz Medical Campus, Aurora, Colorado
  - Local Institution - 2105, Orlando, Florida
  - Local Institution - 2120, Orlando, Florida
  - Children's Healthcare of Atlanta - Egleston Hospital, Atlanta, Georgia
  - Maine Medical Center, Scarborough, Maine
  - Dana Farber Cancer Institute., Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Local Institution - 2110, New Brunswick, New Jersey
  - Local Institution - 2102, New York, New York
  - Levine Children's Hospital- Pediatric Neuro-Oncology, Charlotte, North Carolina
  - Local Institution - 2112, Cleveland, Ohio
  - Local Institution - 2114, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia-Center for Childhood Cancer Research, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - The University of Texas Southwestern Medical Center - Harold C Simmons Comprehensive Cancer Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Local Institution - 2104, Houston, Texas
  - Children's Hospital of Richmond at VCU, Richmond, Virginia
- Australia (4):
  - Local Institution - 6104, Randwick, New South Wales
  - Local Institution - 6103, Westmead, New South Wales
  - Children's Health Queensland Hospital and Health Service, South Brisbane, Queensland
  - Perth Childrens Hospital, Nedlands, Western Australia
- Canada (4):
  - University Of Calgary, Calgary, Alberta
  - Stollery Children'S Hospital, Edmonton, Alberta
  - Children'S Hospital Of Eastern Ontario, Ottawa, Ontario
  - St Justine Hospital, Montreal, Quebec
- Rigshospitalet - Glostrup, Copenhagen, Denmark
- France (10):
  - Local Institution - 6111, Lyon, Rhone
  - Centre Hospitalier Universitaire D'Angers, Angers
  - Centre Hospitalier Universitaire de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Institut d Hematologie et d Oncologie Pediatriques, Lyon
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - Local Institution - 6110, Marseille
  - Local Institution - 6112, Nantes
  - Local Institution - 6109, Paris
  - Institut Gustave-Roussy, Villejuif
  - Local Institution - 6108, Villejuif
- Italy (4):
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Local Institution - 6113, Padua
  - Local Institution - 4302, Rome
  - Local Institution - 6114, Torino
- Singapore (2):
  - National University Hospital, Singapore
  - KK Women's and Children's Hospital, Singapore
- South Korea (4):
  - Local Institution - 6303, Seoul, Seodaemun-gu
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Local Institution - 6304, Seoul
- Spain (11):
  - Hospital Sant Joan De Deu, Esplugues de Llobregat, Barcelona
  - Clínica Universidad de navarra, Pamplona, Navarre
  - Local Institution - 6105, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Local Institution - 6106, Madrid
  - Clinica Universidad de Navarra, Madrid
  - HM Sanchinarro University Hospital, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia
  - Local Institution - 6107, Valencia
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
- United Kingdom (6):
  - Alder Hey Children's NHS Foundation Trust, Liverpool, England
  - Local Institution - 4403, Birmingham
  - University Hospital of Wales, Cardiff
  - Royal Hosp. for Children, Glasgow
  - The Royal Marsden NHS Foundation Trust, London
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data with other researchers.

REFERENCES:
- [Derived] Wachter F, Al-Ibraheemi A, Trissal MC, Hollowell M, DuBois SG, Collins NB, Church AJ, Janeway KA. Molecular Characterization of Inflammatory Tumors Facilitates Initiation of Effective Therapy. Pediatrics. 2021 Dec 1;148(6):e2021050990. doi: 10.1542/peds.2021-050990. PMID 34814185
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04094610.html